CLINICAL TRIAL: NCT05931419
Title: High-Risk prostatE Cancer radiatiOn Versus surgERy (RECOVER)
Brief Title: High-Risk prostatE Cancer radiatiOn Versus surgERy
Acronym: RECOVER
Status: Recruiting | Type: Observational
Sponsor: Comprehensive Cancer Centre The Netherlands (Other)
Responsible Party: Principal Investigator, Berdine Heesterman, Principal Investigator, Comprehensive Cancer Centre The Netherlands
Other Study IDs: 2022-13682
Record Dates: First submitted 2023-04-26; First posted 2023-07-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: Radical prostatectomy; Radiotherapy; Health-related quality of life; Functional outcomes; Progression-free survival; Distant metastases-free survival; Cost-effectiveness
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Robot assisted radical prostatectomy (RARP): Robot-assisted radical prostatectomy, potentially as part of multimodality therapy with adjuvant radiotherapy or with (neo)adjuvant androgen deprivation therapy. Pelvic lymph node dissection (PLND) may be performed for staging purposes. The presence of positive lymph nodes (pN1) upon PLND is not a reason for exclusion and may be followed by adjuvant treatment such as lymph node irradiation.
- External beam radiotherapy (EBRT) combined with androgen deprivation therapy (ADT): External beam radiotherapy (hypofractionated or conventionally fractionated) at a biologically effective dose converted to 2Gy fractions (α/β:1.5) of at least 76Gy. EBRT may be combined with a brachytherapy boost and PLND may be performed for staging purposes. The presence of positive lymph nodes (pN1) upon PLND is not a reason for exclusion and lymph node irradiation may be performed. Patients should receive ADT for at least 6 months.

SUMMARY:
Prospective cohort study comparing robot-assisted radical prostatectomy and external beam radiotherapy combined with androgen deprivation therapy for high-risk non-metastatic prostate cancer in terms of health-related quality of life, functional outcomes, cost-effectiveness, progression-free survival and distant metastasis-free survival.

DETAILED DESCRIPTION:
Detailed description: Robot assisted radical prostatectomy (RARP) and external beam radiotherapy (EBRT) combined with Androgen Deprivation Therapy (ADT) are widely used treatment modalities for high-risk non-metastatic prostate cancer (HR-PCa). Both treatments are associated with adverse effects and can have a great impact on health-related quality of life (HRQoL). To date there is no consensus on which of both is the optimal treatment for men with HR-PCa, as it is unclear which treatment is superior in terms of HRQoL, cost-effectiveness, progression-free survival (PFS) and distant metastases-free survival (DMFS). This is reflected in substantial variation between individual hospitals in the utilization of both treatment options that is not explained by patient- and tumor characteristics or patient preferences. In the RECOVER study we aim to address this knowledge gap. The insights gained can be used to tailor recommendations in (national) guidelines and in shared decision-making tools. This allows healthcare professionals to better inform their patients and allows patients to make well-informed choices.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed de novo non-metastatic high-risk prostate cancer.
* cT3a-bN0M0, according to the 8th edition of the Tumour, Node, Metastasis (TNM) classification, with the exception that clinical T-stage will be based on digital rectal examination and magnetic resonance imaging (the highest stage will be used) and/or
* International Society of Urological Pathology (ISUP) grade ≥4 and/or
* Prostate-Specific Antigen (PSA) value at diagnosis greater than 20 ng/mL
* Fit for treatment with either RARP or EBRT and ADT (WHO performance status 0-1)
* Living in the Netherlands
* Able to read and understand the Dutch language

Exclusion Criteria:

* Histological types other than adenocarcinoma
* Diagnosis and/or treatment in a hospital abroad
* Treatment with Androgen Receptor Targeted Agents (ARTA) as part of the initial treatment plan

Ages: 50 Years to 75 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients with de novo non-metastatic high-risk prostate cancer (cT3a-bN0M0 and/or ISUP grade ≥4 and/or PSA >20ng/ml), who have opted for treatment with RARP or EBRT and ADT and are diagnosed in, or are referred to one of the participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 837 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional outcomes | 3 years after treatment initiation
  Functional outcomes will be measured with the Expanded Prostate Cancer Index Composite Short Form (EPIC-26). The EPIC-26 consists of 5 domains: urinary incontinence, urinary irritation, bowel function, sexual function and hormonal function. Domain scores range from 0-100 (the higher the score the better the function) and the minimally clinically important difference (MCID) per domain is 6-9, 5-7, 4-6, 10-12 and 4-6, respectively.
Health-related quality of life (HRQoL) | 3 years after treatment initiation
  HRQoL will be measured with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30). The questionnaire includes five functional domains (physical, role, cognitive, emotional and social), three symptom domains (fatigue, pain, nausea and vomiting) and a global health/quality of life scale. In addition, there are six separate items assessing dyspnea, insomnia, appetite loss, constipation, diarrhea, and perceived financial impact. For each domain and single item measure, a score from 0 to 100 can be calculated. For the functional domains and the global score, higher scores indicate a higher level of functioning/ better quality of life. In contrast, for the symptom domains and single item measures, a higher score represents a higher level of symptomatology.

SECONDARY OUTCOMES:
Cost-effectiveness | 3 years after treatment initiation
  A cost-utility analysis (CUA) will be conducted from a societal and medical perspective. The societal perspective will specifically focus on the patients out of pocket costs. Utilities will be derived by means of a mapping algorithm for the EORTC QLQ-C30. The derived utility will be used to estimate a Quality adjusted life year (QALY) according to the trapezium rule. Incremental costs between EBRT combined with ADT and RARP will be related to incremental QALYs in a cost-utility ratio (ICUR).
Progression-free survival | 5 years after diagnosis
Distant metastases-free survival | 5 years after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Katja Aben, PhD, Principal Investigator — Comprehensive Cancer Centre The Netherlands; Igle Jan de Jong, MD, PhD, Principal Investigator — University Medical Center Groningen; Floris Pos, MD, PhD, Principal Investigator — Netherlands Cancer Institute/ Antoni van Leeuwenhoek
Locations (29):
- Netherlands (29):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuis Amstelland, Amstelveen
  - Amsterdam UMC, Amsterdam
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - BovenIJ ziekenhuis, Amsterdam
  - OLVG, Amsterdam
  - Wilhelmina Ziekenhuis, Assen
  - Rode Kruis Ziekenhuis, Beverwijk
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Martini ziekenhuis, Groningen
  - Universitair Medisch Centrum Groningen, Groningen
  - Saxenburgh Medisch Centrum, Hardenberg
  - St Jansdal, Harderwijk
  - Spaarne Gasthuis, Hoofddorp
  - Treant, Hoogeveen
  - Dijklander Ziekenhuis, Hoorn
  - Leids Universitair Medisch Centrum, Leiden
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboudumc, Nijmegen
  - Erasmus Medisch Centrum Rotterdam, Rotterdam
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Ommelander Ziekenhuis, Scheemda
  - Haaglanden Medisch Centrum, The Hague
  - Verbeeten Instituut, Tilburg
  - Maxima Medisch Centrum, Veldhoven
  - Zaans Medisch Centrum, Zaandam

REFERENCES:
- [Derived] van der Starre CM, Bangma CH, Bijlsma MJ, van den Bergh ACM, Kiemeney LALM, Kievit W, Vos K, Somford DM, Wildeman SM, Aben KKH, de Jong IJ, Pos FJ, Heesterman BL. External beam radiation therapy versus radical prostatectomy for high-risk prostate cancer: protocol of the RECOVER study. BMC Cancer. 2025 Jan 27;25(1):149. doi: 10.1186/s12885-025-13511-7. PMID 39871169